CLINICAL TRIAL: NCT06937632
Title: Effect of a Nurse-Led Sleep Hygiene Intervention on Sleep Quality Improvement in Elders With Parkinson's Disease: A Quasi-experimental Research Design
Brief Title: Sleep Hygiene Intervention on Sleep Quality Improvement in Elders With Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Rasha salah elsayed eweida, Rasha Eweida, Alexandria University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 4/4/2025
Record Dates: First submitted 2025-04-05; First posted 2025-04-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Sleep Disorder
Keywords: Sleep; Sleep Hygiene; Sleep Quality; Aged; Parkinson's disease; Quasi-Experimental Design
MeSH Terms: conditions — Sleep Wake Disorders; Sleep Hygiene; Sleep Initiation and Maintenance Disorders; Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- interventional group (Experimental): sleep program was done three times a week for 2 weeks for the study group (6 sessions in total). It took roughly 30 minutes for each session. sessions were demonstrated during the first 3 sessions, re-demonstration of all the 3 of other sessions. Over a course of two sessions, the older adults in the intervention group were taught how to perform sleep program. The telephone number of each subject was taken to check their consistency with the proposed nursing interventions.
  Interventions: Behavioral: sleep hygiene intervention

INTERVENTIONS:
Behavioral: sleep hygiene intervention — sleep program was done three times a week for 2 weeks for the study group (6 sessions in total). It took roughly 30 minutes for each session. sessions were demonstrated during the first 3 sessions, re-demonstration of all the 3 of other sessions. Over a course of two sessions, the older adults in the intervention group were taught how to perform sleep program. The telephone number of each subject was taken to check their consistency with the proposed nursing interventions.

SUMMARY:
Sleep disorders (SDs) are one of the most frequent non-motor symptoms of Parkinson's disease (PD), usually increasing in frequency over the course of the disease and disability progression. SDs include nocturnal and diurnal manifestations such as insomnia, REM sleep behavior disorder, and excessive daytime sleepiness. The causes of SDs in PD are numerous, including the neurodegeneration process itself, which can disrupt the networks regulating the sleep-wake cycle and deplete a large number of cerebral amines possibly playing a role in the initiation and maintenance of sleep.

DETAILED DESCRIPTION:
Sleep disorders (SDs) constitute the second most frequent complaint, affecting 64% of PD patients, ranging from 41.1% in naïve patients to 78.3% in complicated patients. SDs in PD are multifactorial and include nocturnal and diurnal manifestations. Reduced sleep efficiency and an increased number of awakenings characterize sleep in PD. These disturbances are linked, on one side, to PD motor (akinesia, rigidity, and dystonia) and autonomic symptoms (nocturia) and, on the other side, to the presence of concomitant SDs such as REM sleep behavior disorder (RBD), restless legs syndrome (RLS), or breathing disorders such as obstructive sleep apnea (OSA). Diurnal manifestations include excessive daytime sleepiness (EDS) and sudden sleep attacks, which could be a consequence of nocturnal sleep impairment or dopaminergic treatment or, more interestingly, to the neurodegenerative process of PD itself dysregulating the circadian sleep-wake rhythm.

ELIGIBILITY:
Inclusion Criteria:

* Elderly individuals aged 60 years or older, with a confirmed diagnosis of Parkinson's Disease.
* Cognitively and physically able to engage in the study.

Exclusion Criteria:

* Participants using sedative medications .

Ages: 58 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 136 (Actual)
Dates: Start 2024-03-12 (Actual); Primary Completion 2024-08-20 (Actual); Study Completion 2024-09-01 (Actual)

PRIMARY OUTCOMES:
The Parkinson's Disease Sleep Scale (PDSS). | 3 month
  The Parkinson's Disease Sleep Scale (PDSS) was developed by (Chaudhuri et al 2002) to assess sleep quality for patients with Parkinson's disease. The scoring system of PDSS scale is:0-30 very poor sleep, 31- 60 poor, 61- 90 neutral, 91- 120 good, 121- 150 very good sleep.

SECONDARY OUTCOMES:
Sleep Hygiene Index (SHI) | 3 month
  Sleep Hygiene Index was developed by (Mastin et al 2006). The Sleep Hygiene Index is a 13 item self-administered index used to assess the presence of behaviors that are thought to compromise sleep quality. The scoring system of (SHI) is: 0-12 very good sleep hygiene, 13- 26 good, 27- 40 poor, 41- 52 very poor sleep hygiene.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Nursing, Alexandria, Egypt